CLINICAL TRIAL: NCT03420014
Title: A Randomized Study Comparing the Efficacy of the Combination of Doxorubicin and the Tumor-targeting Human Antibody-cytokine Fusion Protein L19TNF to Doxorubicin Alone as First-line Therapy in Patients With Metastatic Leiomyosarcoma
Brief Title: Treatment of Metastatic Soft Tissue Sarcoma (STS) Patients (FIBROSARC USA)
Acronym: FIBROSARC US
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Philogen S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PH-L19TNFDOX2-02/17
Record Dates: First submitted 2018-01-12; First posted 2018-02-05 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Leiomyosarcoma
MeSH Terms: conditions — Leiomyosarcoma | interventions — Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Doxorubicin (Active Comparator): Patients will receive a fixed dose doxorubicin, administered as a 15 ± 5 minutes i.v. infusion.
  Interventions: Drug: Doxorubicin
- Arm 2: L19TNF plus doxorubicin (Experimental): Patients will receive a fixed dose of L19TNF in combination with a fixed dose doxorubicin.
  Doxorubicin will be administered as a 15 ± 5 minutes i.v. infusion on day 1 of each 21-day cycle followed by at least 30 minutes pause before starting infusion of L19TNF.
  Interventions: Combination Product: L19TNF plus doxorubicin

INTERVENTIONS:
Drug: Doxorubicin — 75 mg/m2 doxorubicin will be administered once every 3 weeks (Day 1 of every 21-days cycle).
  Arms: Arm 1: Doxorubicin
Combination Product: L19TNF plus doxorubicin — 13 μg/kg L19TNF will be administered on day 1, 3 and 5 of every 21-days cycle in combination with 60 mg/m2 doxorubicin on day 1 of every 21-days cycle.
  Arms: Arm 2: L19TNF plus doxorubicin

SUMMARY:
The present study is an open-label, randomized, controlled, two-arm multi-center study of the efficacy of L19TNF treatment in combination with doxorubicin versus doxorubicin alone in metastatic leiomyosarcoma patients.

DETAILED DESCRIPTION:
In the study, 122 patients will be randomized in a 1:1 ratio to receive doxorubicin treatment (Arm 1) or L19TNF treatment in combination with doxorubicin (Arm 2).

The primary objective of the trial is to evaluate if L19TNF in combination with doxorubicin (Arm 2) given for metastatic leiomyosarcoma improves efficacy measured as progression free survival, as compared to doxorubicin alone (Arm 1).

Anti-cancer activity will be assessed every 6 weeks during therapy and every 12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

Patients may be included in the study if they meet all of the following criteria:

1. Age ≥ 16 years. Patients under 18 years, should be fully grown (proof of fused growth plates).
2. Patients with histological evidence of stage IV metastatic high-grade leiomyosarcoma (grade 2 - 3 according to the Federation Nationale des Centres de Lutte Contre le Cancer (FNCLCC) grading system) not amenable to curative treatment with surgery or radiotherapy.
3. Patients must have at least one unidimensionally measurable lesion by computed tomography as defined by Response Evaluation Criteria In Solid Tumors (RECIST) v.1.1. If only 1 lesion is present at screening this lesion should not have been irradiated during previous treatments.
4. Life expectancy of at least 3 months in the judgment of the investigator.
5. ECOG ≤ 1.
6. Documented negative test for HIV, HBV and HCV. For HBV serology, the determination of HBsAg and anti-HBcAg-Ab is required. In patients with serology documenting previous exposure to HBV, negative serum HBV-DNA is required. For HCV: HCV-RNA or HCV antibody test. Subjects with a positive test for HCV antibody but no detection of HCV-RNA indicating no current infection are eligible.
7. Female patients: negative serum pregnancy test for women of childbearing potential (WOCBP)* within 14 days of starting treatment. WOCBP must agree to use, from the screening to six months following the last study drug administration, highly effective contraception methods, as defined by the "Recommendations for contraception and pregnancy testing in clinical trials" issued by the Head of Medicine Agencies' Clinical Trial Facilitation Group (www.hma.eu/ctfg.html) and which include, for instance, progesterone-only or combined (estrogen- and progesterone-containing) hormonal contraception associated with inhibition of ovulation, intrauterine devices, intrauterine hormone-releasing systems, bilateral tubal occlusion, vasectomized partner or sexual abstinence.
8. Male patients: Male subjects able to father children must agree to use two acceptable methods of contraception throughout the study (e.g., condom with spermicidal gel). Double-barrier contraception is required.
9. Informed consent signed and dated to participate in the study.
10. Willingness and ability to comply with the scheduled visits, treatment plan, laboratory tests and other study procedures.

    * Women of childbearing potential are defined as females who have experienced menarche, are not postmenopausal (12 months with no menses without an alternative medical cause) and are not permanently sterilized (e.g., tubal occlusion, hysterectomy, bilateral oophorectomy or bilateral salpingectomy).

Exclusion Criteria:

Patients will be excluded from participating in this study if they meet one or more of the following criteria:

1. Prior therapy (except surgery and radiation) for unresectable or metastatic malignant soft tissue sarcoma (STS).
2. Patients with primary tumor localized to the extremities and a single resectable synchronous distant metastatic lesion.
3. Patients eligible for neoadjuvant preoperative treatment.
4. Previous treatment with anthracycline-containing chemotherapy.
5. Radiotherapy within 4 weeks prior to start of therapy.
6. Known history of allergy to TNFα, anthracyclines or other intravenously (IV) administered human proteins/peptides/antibodies.
7. Absolute neutrophil count (ANC) < 1.5 x 109/L, platelets < 100 x 109/L and haemoglobin (Hb) < 9.0 g/dl.
8. Chronically impaired renal function as expressed by creatinine clearance < 60 mL/min or serum creatinine > 1.5 ULN.
9. Inadequate liver function (ALT, AST, GGT, ALP or total bilirubin ≥ 1.5 x ULN) or total bilirubin ≥ 1.5 x ULN).
10. International normalized ratio (INR) > 1.5 ULN.
11. Any severe concomitant condition which makes it undesirable for the patient to participate in the study or which could jeopardize compliance with the protocol.
12. History within the last year of cerebrovascular disease and/or acute or subacute coronary syndromes including myocardial infarction, unstable or severe stable angina pectoris.
13. Heart insufficiency (any grade, New York Heart Association (NYHA) criteria).
14. Left Ventricular Ejection Fraction (LVEF) < 50%.
15. Clinically significant cardiac arrhythmias or requiring permanent medication.
16. Abnormalities observed during baseline ECG and Echocardiogram investigations that are considered as clinically significant by the investigator. Subjects with current, or a history of QT/QTc prolongation would be excluded. In particular:

    * patients with a marked prolongation of QT/QTc interval (e.g., repeated demonstration of QTc >480 milliseconds using Fredricia's QT correction formula) are excluded;
    * patients with a history of risk factors for Torsades de Pointes (e.g., heart failure, hypokalemia, family history of prolonged QT syndrome) are excluded;
    * patients who require the use of concomitant medications that prolong the QT/QTc interval are excluded.
17. Uncontrolled hypertension, despite optimal therapy.
18. Ischemic peripheral vascular disease (Grade IIb-IV according to Leriche-Fontaine classification).
19. Severe diabetic retinopathy such as severe non-proliferative retinopathy and proliferative retinopathy.
20. Major trauma including major surgery (such as abdominal/cardiac/thoracic surgery) within 4 weeks of administration of study treatment.
21. Pregnancy or breast-feeding.
22. Requirement of chronic administration of corticosteroids or other immunosuppressant drugs. Limited use of corticosteroids to treat or prevent acute hypersensitivity reactions is not considered an exclusion criterion.
23. Presence of active and uncontrolled infections or other severe concurrent disease, which, in the opinion of the investigator, would place the patient at undue risk or interfere with the study.
24. Known active or latent tuberculosis (TB).
25. Concurrent malignancies other than soft tissue sarcoma (STS), unless the patient has been disease-free for at least 2 years.
26. Growth factors or immunomodulatory agents within 7 days prior to the administration of study treatment.
27. Serious, non-healing wound, ulcer or bone fracture.
28. Allergy to study medication or excipients in study medication.
29. Concurrent therapy with anticoagulants.
30. Concurrent use of other anti-cancer treatments or agents other than study medication.
31. Any recent live vaccination within 4 weeks prior to treatment or plan to receive vaccination during the study.

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2018-12-27 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | From randomization up to week 72
  Progression-free survival PFS in a time-to-event analysis in the L19TNF plus Doxorubicin control group (Arm 2) versus the Doxorubicin alone treatment group (Arm 1).

SECONDARY OUTCOMES:
Overall survival (OS) | From week 1 up to week 72, every 6 weeks; from week 73 up to week 144, every 12 weeks;
  Overall survival (OS) in the L19TNF plus Doxorubicin treatment group (Arm 2) versus Doxorubicin alone (Arm 1) will be evaluated in time to event analysis.
Overall response rate (ORR) | 1) From week 1 up to week 18, every 6 weeks; 2) from week 19 up to week 72, every 12 weeks (Maintenance); 3) EoT: at week 22/23 (only Induction) and at week 72 (Maintenance); 4) Follow-up: from week 22/23 (EoT) up to week 72, every 12 weeks.
  Overall Response Rate (ORR) assessed by BIRC, i.e. rate of CR and PR of L19TNF plus Doxorubicin treatment group (Arm 2) versus Doxorubicin alone (Arm 1).
Duration of response (DOR) | 1) From week 1 up to week 18, every 6 weeks; 2) from week 19 up to week 72, every 12 weeks (Maintenance); 3) EoT: at week 22/23 (only Induction) and at week 72 (Maintenance); 4) Follow-up: from week 22/23 (EoT) up to week 72, every 12 weeks.
  Duration of Response (DOR) assessed by BIRC in the L19TNF plus Doxorubicin treatment group (Arm 2) versus Doxorubicin alone (Arm 1).
Progression-free survival (PFS) rate | 1) From week 1 up to week 18, every 6 weeks; 2) from week 19 up to week 72, every 12 weeks (Maintenance); 3) EoT: at week 22/23 (only Induction) and at week 72 (Maintenance); 4) Follow-up: from week 22/23 (EoT) up to week 72, every 12 weeks.
  PFS rate of L19TNF plus Doxorubicin treatment group (Arm 2) versus Doxorubicin alone (Arm 1).
Overall survival (OS) rates | From week 1 up to week 144.
  Overall survival (OS) rates in the L19TNF plus Doxorubicin treatment group (Arm 2) versus Doxorubicin alone (Arm 1).
Number of patients with adverse events (AEs). | From week 1 up to week 72.
Percentage of participants with worst on-study hematological and chemistry abnormalities. | From week 1 up to week 72.
Percentage of participants with Electrocardiogram (ECG) and Echocardiogram (ECHO) abnormality findings. | From week 1 up to week 72, every 6 weeks.
Number of Participants With Clinically Significant Abnormalities in Vital Signs (Systolic and Diastolic Blood Pressure, Temperature, Heart Rate). | From week 1 up to week 72.
Number of Participants With Clinically Significant Physical Examination Abnormalities (General Appearance, Skin, Eyes, Ears-Nose-Throat, Breast, Head and Neck, Lungs, Heart, Abdomen, Lymph Nodes, Musculoskeletal) | From week 1 up to week 72.
Human anti-fusion protein antibodies (HAFA) levels against L19TNF. | At day 1 of week 1 and week 2; at day 1 from week 4 up to week 18, every 3 weeks; at week 22-23 (EoT); at week 23-24 (first follow-up visit)
Maximum drug concentration [Cmax]. | At day 1, 2 ,3 and 5 of week 1
  Pharmacokinetics assessment of L19TNF through blood sampling.
Time to reach maximum drug concentration [Tmax]. | At day 1, 2 ,3 and 5 of week 1
  Pharmacokinetics assessment of L19TNF through blood sampling.
Terminal half-life [t1/2]. | At day 1, 2 ,3 and 5 of week 1
  Pharmacokinetics assessment of L19TNF through blood sampling.
Area under the drug concentration-time curve, extrapolated to infinity [AUC]. | At day 1, 2 ,3 and 5 of week 1
  Pharmacokinetics assessment of L19TNF through blood sampling.
Maximum drug concentration [Cmax]. | At day 1, 2 ,3 and 5 of week 1
  Pharmacokinetics assessment of doxorubicin through blood sampling.
Time to reach maximum drug concentration [Tmax]. | At day 1, 2 ,3 and 5 of week 1
  Pharmacokinetics assessment of doxorubicin through blood sampling.
Terminal half-life [t1/2]. | At day 1, 2 ,3 and 5 of week 1
  Pharmacokinetics assessment of doxorubicin through blood sampling.
Area under the drug concentration-time curve, extrapolated to infinity [AUC]. | At day 1, 2 ,3 and 5 of week 1
  Pharmacokinetics assessment of doxorubicin through blood sampling.

CONTACTS AND LOCATIONS:
Overall Officials: Scott H. Okuno, M.D., Principal Investigator — Mayo Clinic, Rochester, MN
Locations (8):
- United States (8):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Sarcoma Oncology Research Center (SORC) Cancer Center of Southern California, Santa Monica, California
  - Mayo Clinic Hospital, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Rutgers Cancer Institute of New Jersey 195 Little Albany Street New Brunswick, NJ 08901 Room 2031, New Brunswick, New Jersey
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Seattle Cancer Care Alliance 825 Eastlake Ave. E. Seattle, WA 98109 Mail Stop CE2-128, Seattle, Washington